CLINICAL TRIAL: NCT05967429
Title: Predictors of Sorafenib Response in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Predictors of Sorafenib Response in HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-23-07-07PD
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Nutrition assessment; HCC; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatocellular carcinoma receiving sorafenib: Patient with advanced stage HCC receiving sorafenib
  Interventions: Diagnostic Test: The neutrophil-to- lymphocyte ratio; Diagnostic Test: Prognostic nutrition index

INTERVENTIONS:
Diagnostic Test: The neutrophil-to- lymphocyte ratio — It was calculated by dividing the neutrophil count by the lymphocyte count.
  Other Names: NLR
Diagnostic Test: Prognostic nutrition index — It was calculated using the following formula: serum albumin (g/L) + 0.005 × total lymphocyte count/μL
  Other Names: PNI

SUMMARY:
Evaluating the nutrition status of patients with advanced HCC who received sorafenib.

Using the pretreatment nutrition status and quality of life as predictors to sorafenib response

DETAILED DESCRIPTION:
This a cross sectional study will be conducted on 100 HCC treated with sorafenib Data were gathered from medical records, including

age sex body weight and height (BMI) pre-therapy laboratory counts of white cells, neutrophils, lymphocytes, monocyte, hemoglobin and platelets; bilirubin, albumin and globulin concentration, AST, ALT, AFP, PT and CONC

Barcelona Clinic Liver Cancer Stage (BCLC) of all patients

The neutrophil-to- lymphocyte ratio (NLR) was calculated by dividing the neutrophil count by the lymphocyte count.

The platelet- to-lymphocyte ratio (PLR) was calculated by dividing the platelet count by the lymphocyte count.

Weight loss difference after treatment Portal hypertension was defined as presence of either collaterals on radiological examination, esophageal varices by upper gastrointestinal endoscopy and/or thrombocytopenia.

Quality of life assessment. QoL was assessed using FACT Hepatobiliary Symptom Index (FHSI-8) Questionnaire. QoL was assessed at base line and 3-6 months after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCC recieved sorafenib

Exclusion Criteria:

* Patient refuse to participate
* Patients recieving other treatment modalities

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hepatocellular carcinoma patient receiving sorafenib
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
assessment of nutrition status | Augest 2023 to March 2024
  Prognostic nutrition index
Predictors of sorafenib response | Augest 2023 to March 2024
  The neutrophil-to- lymphocyte ratio
Assess the quality of life | Augest 2023 to March 2024
  using FACT Hepatobiliary Symptom Index

CONTACTS AND LOCATIONS:
Overall Officials: Amr Zagloul, MD, Study Director — Sohag University; Ahmed othman, MD, Study Chair — Sohag University; Rafat Abd El Aal, MD, Study Chair — Sohag University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takagi K, Buettner S, Ijzermans JNM. Prognostic significance of the controlling nutritional status (CONUT) score in patients with colorectal cancer: A systematic review and meta-analysis. Int J Surg. 2020 Jun;78:91-96. doi: 10.1016/j.ijsu.2020.04.046. Epub 2020 Apr 23. PMID 32335238